CLINICAL TRIAL: NCT01718548
Title: The Effects of Cordyceps Sinensis and Lingzhi on Cardiovascular Fitness and Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0062-12-HYMC
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Physical Fitness; Executive Function
MeSH Terms: interventions — Tea; Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CS and Lingzhi (Active Comparator): CS liquid (each dosage is a bottle of liquid containing 30 ml: comprising 75% of CS, 6% Lingzhi, 6% shitake, 5% bamboo shoot, 2% honey, 0.1% potassium sorbet and 5.9% pure water) and Lingzhi capsule (each capsule contains 620mg of: 52.42% Lingzhi, 28.23% CS, and 19.35% soy gel ) ; one quarter bottle of CS to be ingested twice a day, and the Lingzhi capsule to be taken once a day, both for a period of 28 days.
  Interventions: Dietary Supplement: Cordyceps Sinensis (CS) and Lingzhi
- Placebo (Placebo Comparator): Liquid tea ingested twice a day and flour-filled capsules ingested once a day over a period of 28 days
  Interventions: Dietary Supplement: Tea and Flour

INTERVENTIONS:
Dietary Supplement: Cordyceps Sinensis (CS) and Lingzhi
  Arms: CS and Lingzhi
Dietary Supplement: Tea and Flour — Placebo
  Arms: Placebo

SUMMARY:
Cordyceps Sinensis (CS) and Lingzhi extracts have been used in Chinese Medicine for many years for treatment of a variety of conditions. The aim of this study is to evaluate the effects of oral ingestion of CS and Lingzhi extracts of a period of 28 days on cardiopulmonary fitness and cognitive functioning in young, healthy physical education students.

ELIGIBILITY:
Inclusion Criteria:

* Physical education students

Exclusion Criteria:

* All others

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Cardiopulmonary Fitness after Ingestion of CS and Lingzhi Extracts | 28 days
  Before and after 28-day ingestion of CS and Lingzhi extracts, subjects will undergo a graded exercise test on a treadmill and results will be compared.

OTHER OUTCOMES:
Effect of CS and Lingzhi on Cognitive Functioning | 28 days
  Before and after 28-day ingestion of CS and Lingzhi the subjects undergo computerized cognitive tests and results will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Wingate Institute, Netanya, Israel